CLINICAL TRIAL: NCT02721264
Title: Fecal Microbiota Therapy Versus Standard Therapy in NASH Related Cirrhosis: A Randomized Control Trial
Brief Title: Fecal Microbiota Therapy Versus Standard Therapy in NASH Related Cirrhosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-NASH-03
Record Dates: First submitted 2016-03-01; First posted 2016-03-29 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fecal Microbiota Transplantation (FMT) (Experimental): The recipient will receive healthy donor, prepared fecal installations through a Naso-gastric tube, 100 ml once a month for 5 month.
  Interventions: Biological: Fecal Microbiota Transplant
- Standard Treatment Care (Active Comparator)
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Biological: Fecal Microbiota Transplant
  Arms: Fecal Microbiota Transplantation (FMT)
Other: Standard Medical Treatment
  Arms: Standard Treatment Care

SUMMARY:
Patients of NASH (Non Alcoholic Steatohepatitis) cirrhosis with current or prior histological evidence of steatosis or steatohepatitis admitted under the Department of Hepatology at Institute of Liver and Biliary Sciences, who meet the inclusion criteria and who provide informed consent will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age more then 18 years.
2. All patients with cirrhosis with current or previous histological evidence of steatosis or steatohepatitis.
3. Histologic evidence of definite or probable NASH based upon a liver biopsy prior to enrollment and a NAFLD activity score (NAS) ≥5 with ≥1 in each component of the NAS score (steatosis, scored 0-3, ballooning degeneration, 0-2, and lobular inflammation, 0-3).
4. No past history of upper GI bleeding, ascites, hepatic encephalopathy

Exclusion Criteria:

1. Diagnosis of liver disease other than NASH cirrhosis
2. History of gastrointestinal bleeding, ascites, hepatic encephalopathy
3. Ongoing bacterial infection requiring antibiotic treatment.
4. Current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening
5. Treatment with antibiotics or probiotics in the preceding 3 months.
6. Inability to safely obtain a liver biopsy or perform an upper GI endoscopy
7. Psychiatric disorder
8. HIV
9. Pregnant women
10. Patients on SBP (Spontaneous Bacterial Peritonitis) prophylaxis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Hepatic Venous Pressure Gradient in the two groups from baseline. | 1 year

SECONDARY OUTCOMES:
Improvement in liver function test as compared to baseline. | 1 year
  Improvement is defined as Serum bilirubin,AST,ALT,serum Albumin within normal limits
Improvement in Liver Stiffness Measurement as compared to baseline. | 1 year
  LSM < 10 Kpa
Assess improvement in insulin resistance (Fasting plasma and insulin levels, HOMA-IR) | 1 year
  HOMA IR <2.5
Incidence of new onset upper gastrointestinal bleed in both groups | 1 year
development of new onset of ascites in both groups. | 1 year
Number of Spontaneous Bacterial peritonitis cases in both groups. | 1 year
ACLF (Acute on Chronic Liver failure) cases in both groups. | 1 year
Reduction in hepatic and systemic inflammatory markers like TNF-α in both groups | 1 year
Reduction in hepatic and systemic inflammatory markers like C Reactive Protein in both groups | 1 year
Reduction in hepatic and systemic inflammatory markers like serum endotoxins in both groups. | 1 year
Histological and permeability changes in the duodenal biopsy in both groups. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr Abhinav Verma, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aghara H, Patel M, Chadha P, Parwani K, Chaturvedi R, Mandal P. Unraveling the Gut-Liver-Brain Axis: Microbiome, Inflammation, and Emerging Therapeutic Approaches. Mediators Inflamm. 2025 Jun 18;2025:6733477. doi: 10.1155/mi/6733477. eCollection 2025. PMID 40568349